CLINICAL TRIAL: NCT04763863
Title: The Nordic Consensus Study
Acronym: NCS
Status: Completed | Type: Observational
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: CP339
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Stoma Site Leakage; Quality of Life; Nurse's Role; Stoma Ileostomy; Colostomy Stoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ostomates: Ostomates with leakage issues and stoma created at least 3 months ago
  Interventions: Other: Body Assessment Tool
- Stoma care nurses: Stoma care nurses from Denmark, Finland, Norway and Sweden who had agreed to participate. Invitations were sent to stoma care nurses randomly selected from among those working in relatively large stoma care clinics.
  Interventions: Other: Clinical usability evaluation of the Body Assessment Tool

INTERVENTIONS:
Other: Body Assessment Tool — Assessment tool to evaluate stoma to find proper ostomy products
  Groups: Ostomates
Other: Clinical usability evaluation of the Body Assessment Tool — The stoma care nurses evaluated the clinical usability of the Body Assessment Tool, which included answering the following questions:
  Does the tool offer value in clinical practice? Does it provide a good starting point when choosing ostomy product(s)? Does it help raise the quality of care? Participants provided their responses on a 6 point-scale (1-6), where 1 indicated the lowest satisfaction and 6 the greatest satisfaction with the tool.
  Groups: Stoma care nurses

SUMMARY:
A Body Assessment Tool was developed to provide nurses with a more structured approach when choosing ostomy products. The Body Assessment Tool will to be evaluated in clinical settings.

DETAILED DESCRIPTION:
The primary objective is to evaluate the usability of the Body Assessment Tool for the nurse. The secondary objectives are to explore if the use of Body Assessment Tool has an impact on the leakage associated Quality of Life and leakage incidences for individuals living with ostomies.

Forty to fifty ostomates will be enrolled from each Nordic country (i.e. Denmark, Sweden, Norway and Finland). The users will be recruited from 5-10 clinics in each country. The evaluation will include 1 visit at the clinic and at least 1 phone call visit to the user (end-of study phone visit).

The usability of the Body Assessment Tool will be evaluated by the nurses. The user's leakage and QoL will be evaluated by the end-users.

ELIGIBILITY:
Inclusion Criteria:

* Ostomates
* Male or female ≥18years
* Leakage issues

Exclusion Criteria:

* Requires a caretaker or is unable to participate in the study
* Is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ostomates with leakage problems in need for stoma care
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Coloplast Denmark A/s, Humlebæk, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Stoma Care Nurses: Stoma care nurses from Denmark, Finland, Norway and Sweden who had agreed to participate.
Period: Overall Study
Arm/Group | Ostomates | Stoma Care Nurses
Started | 99 | 22
Completed | 68 | 22
Not Completed | 31 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nurse: Stoma care nurses from Denmark, Finland, Norway and Sweden who had agreed to participate.
- Total: Total of all reporting groups
Arm/Group | Ostomates | Nurse | Total
Number analyzed (Participants) | 68 | 22 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Stoma care nurses performed an evaluation of the clinical usability of the Body Assessment Tool on the Ostomates and baseline characteristics for the nurses themselves was therefore not collected.
  years
    number analyzed (Participants) | 68 | 0 | 68
    (all) | 67.8 (12.1) |  | 67.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants had missing data in Ostomates group
  Stoma care nurses performed an evaluation of the clinical usability of the Body Assessment Tool on the Ostomates and baseline characteristics for the nurses themselves was therefore not collected.
  Participants
    number analyzed (Participants) | 66 | 0 | 66
    Female | 40 |  | 40
    Male | 26 |  | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Population: Stoma care nurses performed an evaluation of the clinical usability of the Body Assessment Tool on the Ostomates and baseline characteristics for the nurses themselves was therefore not collected.
  participants
    Denmark: number analyzed (Participants) | 68 | 0 | 68
    Denmark | 29 |  | 29
    Sweden: number analyzed (Participants) | 68 | 0 | 68
    Sweden | 8 |  | 8
    Norway: number analyzed (Participants) | 68 | 0 | 68
    Norway | 19 |  | 19
    Finland: number analyzed (Participants) | 68 | 0 | 68
    Finland | 12 |  | 12
Type of ostomy [Count of Participants; unit: Participants] — Population: 1 individual with missing data in Ostomates group
  Stoma care nurses performed an evaluation of the clinical usability of the Body Assessment Tool on the Ostomates and baseline characteristics for the nurses themselves was therefore not collected.
  Participants
    number analyzed (Participants) | 67 | 0 | 67
    Colostomy | 32 |  | 32
    Ileostomy | 25 |  | 25
    Urostomy | 10 |  | 10
Consistency of output [Count of Participants; unit: Participants] — Population: 4 individuals with missing data in Ostomates group
  Stoma care nurses performed an evaluation of the clinical usability of the Body Assessment Tool on the Ostomates and baseline characteristics for the nurses themselves was therefore not collected.
  Participants
    Thick stool: number analyzed (Participants) | 64 | 0 | 64
    Thick stool | 25 |  | 25
    Liquid stool: number analyzed (Participants) | 68 | 0 | 68
    Liquid stool | 29 |  | 29
    Urine: number analyzed (Participants) | 68 | 0 | 68
    Urine | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Body Assessment Tool Based on the Nurse Evaluation Form
Description: Clinical usability evaluation of the Body Assessment Tool was based on a 6-point scale (1 being lowest satisfaction - 6 being highest satisfaction) in response to the three questions: "Does the tool offer value in clinical practice?", "Does it provide a good starting point when choosing ostomy product(s)?", and "Does it help raise the quality of care?".
Time Frame: Visit 2: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stoma Care Nurses
Number analyzed (Participants) | 22
score on a scale
  Does the tool offer value in clinical practice? | 4.6 (1.1)
  Does it provide a good starting point when choosing ostomy product(s)? | 5.1 (0.8)
  Does it help raise the quality of care? | 4.7 (1.3)

2. Secondary Outcome: QoL (Based on the Three OLI Domain Scores (Emotional Impact, Usual and Social Activities, and Coping and in Control)
Description: The Ostomy Leak Impact (OLI) score comprises 22 questions, divided into the three domains: emotional impact (10 questions), usual and social activities (8 questions), and coping and in control (4 questions). The response to each question is rated on a 4-point Likert scale: 'all of the time', 'often', 'sometimes', and 'rarely or never' with higher scores indicating a better outcome. These responses are scored 0,1,2, and 3 respectively in the data processing. Because the domains contain a different number of questions, the score for each was transformed to the range of 0-100 to enable comparison across the three domains; the higher the score, the better level of leakage-related quality of life.
Time Frame: Visit 1 (Week 0) and Visit 2 (Week 4)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ostomates
Number analyzed (Participants) | 68
score on a scale
  emotional impact Visit 1 | 62.1 [56.1 to 68.1]
  emotional impact Visit 2 | 80.0 [74.1 to 86.0]
  usual and social activities Visit 1 | 78.5 [73.1 to 83.8]
  usual and social activities Visit 2 | 89.2 [83.6 to 94.7]
  coping and in control Visit 1 | 67.3 [60.8 to 73.7]
  coping and in control Visit 2 | 83.5 [77.0 to 89.9]

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Ostomates
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT04763863/Prot_SAP_000.pdf